CLINICAL TRIAL: NCT02571023
Title: Multicenter Clinical Study on Diagnosis and Treatment of Skull Base Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hou Lijun (Other)
Responsible Party: Sponsor-Investigator, Hou Lijun, Director of Neurosurgery Department, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Other Study IDs: Skull Base Trauma 2016
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Skull Injury Trauma
Keywords: Skull Base Trauma; microscope surgery; neuroendoscope surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: microscope surgery
Procedure: neuroendoscope surgery

SUMMARY:
The purposes of this study are as follows:

1. to collect the largest epidemiological data of skull base trauma and analyze the related influence factors of mortality and morbidity.
2. to establish a set of standard classification methods of skull base trauma and to establish a standard rating scale for each type of trauma.
3. to select optimized conservative and surgical treatments of skull base trauma and to compare the therapeutic effect between microscope surgery and neuroendoscopic surgery.
4. to clear the epidemiological characteristics of the skull base trauma combined with paroxysmal sympathetic hyperactivity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Skull Base Trauma

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with skull base trauma in inpatient ward.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
mortality | 1 year
disability rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Hou, MD, Study Chair — Department of Neurosurgery, Shanghai Changzheng Hospital
Locations (1):
- Department of Neurosurgery, Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China